CLINICAL TRIAL: NCT04001777
Title: A Phase Ib Study of Safety and Efficacy of APG-1252 in Combination With Osimertinib (AZD9291) in EGFR TKI Resistant NSCLC Patients
Brief Title: A Study of APG-1252 Plus Osimertinib(AZD9291) in EGFR TKI Resistant NSCLC Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG1252NC101
Record Dates: First submitted 2019-06-20; First posted 2019-06-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer
MeSH Terms: interventions — pelcitoclax; Injections; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- APG-1252 plus Osimertinib (AZD9291) (Experimental): APG-1252 will be explored sequentially using a standard 3+3 escalation scheme at the dose escalation phase; Dose of osimertinib will be fixed at 80mg QD based on approved label.
  Interventions: Drug: APG-1252; Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: APG-1252 — Multiple dose cohorts, 30 minute IV infusion, weekly for 3 weeks of a cycle with 21days.
  Other Names: APG-1252 for injection
Drug: Osimertinib Mesylate Tablets — Osimertinib Mesylate Tablets 40mg/80 mg, one time a day until disease progression
  Other Names: AZD9291

SUMMARY:
There are unmet medical needs in patients who resist to EGFR TKIs, especially to osimertinib; APG-1252 shows synergy with osimertinib in both osimertinib treatment naïve and resistant cell lines. This study is to explore the safety and efficacy of the combination of APG-1252 and osimertinib in 3rd generation TKI resistant patients and 3rd generation TKI treatment naïve patients.

DETAILED DESCRIPTION:
This is an open-label, single-arm, multicenter, phase 1b study and consists of two stages: dose finding and dose expansion.

The dose-finding stage will explore the safety and tolerability of APG-1252 at different dose levels combined with osimertinib mesylate tablets (hereinafter referred to as osimertinib) at a fixed dose level and determine the MTD and/or RP2D of APG-1252. According to the results from the ongoing phase 1 clinical trials (APG-1252-US-001, APG-1252-AU-001, APG-1252-CH-001) of APG-1252 currently, the starting dose of APG-1252 is set as 240 mg in the study. The 3+3 design will be implemented. The dose for successive cohorts will be escalated to 320 mg and 400 mg or de-escalated to 160 mg and 80 mg based on the safety of the starting dose.

During the dose-expansion period, the efficacy of APG-1252 combined with osimertinib will first be studied in patients with NSCLC that has progressed after treatment with third-generation EGFR TKIs. There will be a total of 20 subjects in Cohort 1. If at least one of the first 10 evaluable patients achieves a response (confirmed complete response [CR] or partial response [PR], assessed by the investigator as per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) in the dose-expansion period, Cohort 2 and Cohort 3 will be initiated at the same time.

ELIGIBILITY:
Inclusion Criteria:

Only applicable to the dose-finding stage:

Patients with NSCLC with disease progression after first-line EGFR TKI and platinum-based chemotherapy.

Only applicable to dose-expansion stage:

Cohort 1: Patients with NSCLC with disease progression after third-generation EGFR TKI and platinum-based chemotherapy.

Cohort 2: Patients with NSCLC with disease progression after first- or second-generation EGFR TKI and platinum-based chemotherapy.

Cohort 3: Patients with advanced EGFR-mutated NSCLC not previously treated with TKI.

Applicable to any phase:

1. Histologically or cytologically confirmed incurable advanced or metastatic non-small cell lung cancer.
2. At least 1 measurable lesion (RECIST 1.1).
3. Confirmed EGFR mutation positive before start use prior EGFR TKI(s) .
4. Willing to biopsy or to supply achieved tumor sample which biopsy after the most recent treatment.
5. Male or female patients age ≥18 years.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
7. Estimated OS ≥3 months.
8. Adequate hematologic and bone marrow functions.
9. Adequate renal and liver function.
10. Brain metastases with clinically controlled neurologic symptoms.
11. Had recovered from all toxicities related to prior anticancer therapies to grade ≤ 2, except for patients with grade 2 nausea/vomiting and/or grade 2 diarrhea despite optimal supportive therapy who will not be allowed to participate in the study.
12. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential (postmenopausal women must have been amenorrhea for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug.
13. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).
14. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Received chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy (hormones for hypothyroidism or estrogen replacement therapy (ERT), anti-estrogen analogs, agonists required to suppress serum testosterone levels are permitted); or any investigational therapy; , or has had tumor embolization or tumor lysis syndrome (TLS) within 28 days prior to the first dose of study drug.
2. Received TKIs targeted therapy (except third generation EGFR TKIs) within 14 days prior to the first dose of study drug.
3. A history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, or any evidence of clinically active interstitial lung disease.
4. Any of the following cardiac criteria: screening period resting period QTC > 470 milliseconds (clinical electrocardiograph report value; if a single time> 470 milliseconds, take the average of 3 inspections); rhythm of resting electrocardiogram (ECG), any clinically important abnormality of conduction or morphology (e.g., complete left bundle branch block, Grade 3 heart block, Grade 2 heart block); family history of congenital long QT prolongation syndrome or long QT syndrome.
5. Evidence of any serious or uncontrolled systemic disease; various chronic active infections such as hepatitis B (HBV-DNA ≥ 104 copy number/ml or 2000 IU/ml), hepatitis C and HIV; uncontrollable Hypertensive patients (requires 2 or more drugs to control blood pressure); unstable angina; angina pectoris within 3 months prior to study; congestive heart failure (NYHA class II or higher); myocardial infarction (NSTEMI or STEMI) history in 6 months before study enrollment; severe arrhythmia requiring medical attention; severe liver, kidney, gastrointestinal or metabolic diseases.
6. Patients who are unable to stop taking drugs or herbal medicine that are strong inhibitors or inducers of CYP3A within 1 week before the first study drug administration and during the treatment. However, patients who discontinue use of these compounds at least 1 week prior to receiving this regimen are eligible.
7. Hemorrhagic constitution/disease, such as a history of non-chemotherapy-induced thrombocytopenic hemorrhage or a history of ineffective platelet transfusion within 1 year prior to the first dose of study drug; Severe gastrointestinal bleeding occurred within 3 months prior to the first dose of study drug; Active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AIHA), etc.
8. Use a therapeutic dose of anticoagulant or antiplatelet agent before the first use of APG-1252 or within 7 days of central catheter placement (if platelet count is stable (≧50×109/L), Subjects who previously received aspirin to prevent thrombosis therapy can reuse low-dose aspirin (i.e., up to 100 mg QD) after 3 weeks of study drug treatment; Decisions regarding anticoagulants and antiplatelet therapy will be determined by the investigator and the sponsor; Allow low-dose anticoagulant drugs to maintain central venous catheters open.
9. Received a biologic (G-CSF, GM-CSF or erythropoietin) within 28 days prior to the first dose of study drug.
10. According to the investigator's judgment, patients who did not fully recover after surgery. Patients who underwent major surgery within 28 days prior to the first study drug and who underwent minor surgery within 7 days prior to the start of the study.
11. Other malignancies have been diagnosed within 5 years prior to the first use of the study drug; except effectively treated skin basal cell carcinoma, cutaneous squamous cell carcinoma, and/or effectively resected orthotopic cervical cancer and/or breast cancer.
12. Female patients during pregnancy or lactation.
13. Previous allergies or intolerance to treatment with osimertinib.
14. A diagnosis of febrile neutropenia within one week prior to the first use of the study drug.
15. Prior treatment with Bcl-2/Bcl-xL inhibitors.
16. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days
  To determine the maximum tolerated dose (MTD) of APG-1252 in subjects with NSCLC
Recommended Phase 2 dose (RP2D) | 21 days
  Recommended Phase 2 dose (RP2D) of APG-1252 in subjects with NSCLC

SECONDARY OUTCOMES:
efficacy assessment: Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | Every 6 weeks up to 2 years
  To assess efficacy in subjects with NSCLC using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Professor, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - Sun-Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Provincial people's Hospital, Zhengzhou, Henan
  - First Hospital of Jilin University, Changchun, Jilin
  - Jilin Provincial Cancer Hospital, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No